CLINICAL TRIAL: NCT06809413
Title: Clinical Study on the Early Bactericidal Activity of Sitafloxacin Against Mycobacterium Abscessus Disease
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Nie WenJuan, chief physician, Beijing Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCP-TB-2025-1-28
Record Dates: First submitted 2025-01-28; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Fluoroquinolone; Mycobacterium
Keywords: Mycobacterium abscessus; Sitafloxacin; early bactericidal activity; Colony forming units; time to positivity
MeSH Terms: conditions — Mycobacterium Infections; Mycobacterium Infections, Nontuberculous | interventions — sitafloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sitafloxacin group (Experimental): This study intends to enroll 12 patients with Mycobacterium abscessus infections. They will be administered sitafloxacin continuously for 14 days, and sputum samples will be collected for colony-forming units counting and time to positivity observation to evaluate the efficacy of the antibacterial agent.
  Study Medication: Sitafloxacin 100mg once daily for 14 days.
  Interventions: Drug: Sitafloxacin

INTERVENTIONS:
Drug: Sitafloxacin — Study medication: Sitafloxacin 100mg QD for 14 days.

SUMMARY:
This study is a single-center, open-label clinical trial designed to evaluate the early bactericidal activity (EBA) of sitafloxacin against Mycobacterium abscessus disease. Patients with Mycobacterium abscessus disease were enrolled and treated with sitafloxacin monotherapy for 14 days. Colony forming units (CFU) and time to positivity (TTP) in sputum cultures were analyzed and compared. By assessing the impact of sitafloxacin monotherapy on the bacteria in the sputum of patients with Mycobacterium abscessus disease, the early bactericidal activity of sitafloxacin was evaluated, providing a basis for the selection of new drugs for the treatment of Mycobacterium abscessus disease.

DETAILED DESCRIPTION:
This study is a single-center, open-label clinical trial designed to evaluate the early bactericidal activity (EBA) of sitafloxacin against Mycobacterium abscessus disease. Patients with Mycobacterium abscessus disease were enrolled and treated with sitafloxacin monotherapy for 14 days. Colony forming units (CFU) and time to positivity (TTP) in sputum cultures were analyzed and compared. By assessing the impact of sitafloxacin monotherapy on the bacteria in the sputum of patients with Mycobacterium abscessus disease, the early bactericidal activity of sitafloxacin was evaluated, providing a basis for the selection of new drugs for the treatment of Mycobacterium abscessus disease.

Study medication: Sitafloxacin 100mg QD for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* (1) Diagnosed or clinically diagnosed with Mycobacterium abscessus pulmonary disease within 6 months prior to enrollment; (2) Voluntarily participate in this study and sign the informed consent form; (3) Agree to use contraception voluntarily.

Exclusion Criteria:

* (1) Received glucocorticoids or immunosuppressants within 90 days prior to enrollment; (2) Pregnant women or postpartum lactating women; (3) Patients with evidence of fluoroquinolone resistance or allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Early bactericidal activity | 14 days
  Patients with Mycobacterium abscessus infections were enrolled and treated with sitafloxacin monotherapy for 14 days to assess its early bactericidal activity. This involved analyzing and comparing the colony-forming units and time to positivity in sputum cultures to evaluate the impact of sitafloxacin on the bacteria in the sputum of patients with Mycobacterium abscessus infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing chest hospital affiliated to Capital medical university, Beijing Tuberculosis & Thoracic Tumor Research Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
In our hospital, researchers are not allowed to upload patient data or hospital information to websites without authorization.